CLINICAL TRIAL: NCT07219264
Title: Mental Health CPR: Transforming Cancer Survivors' Mental Health With Community Participatory Reach
Brief Title: Mental Health CPR for Cancer Survivors
Acronym: MH-CPR CaS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: University of Rochester (Other); University of Puerto Rico Medical Sciences Campus (Unknown)
Responsible Party: Principal Investigator, Eida M Castro-Figueroa, Principal Investigator, Ponce Medical School Foundation, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01CA290613 (NIH)
Record Dates: First submitted 2025-10-15; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Mental Health Care; Mental Health; Depression Anxiety Disorder
Keywords: Mental Health; Distress; Depression; Anxiety
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Although participants and intervention facilitators are aware of group assignment due to the behavioral nature of the intervention, masking is applied to the outcomes assessment process. Laboratory personnel responsible for the processing and analysis of saliva samples for biological markers are blinded to group assignment to maintain objectivity in outcome measurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health CPR Intervention (Experimental): Participants in this arm will receive the Mental Health PR community-based behavioral intervention. The program consist pf structured sections facilitated by trained Community Mental Health Workers (CHMWs) focused on improving communication, stress management, and access to mental health services. Sessions are delivered in small groups through culturally tailored materials and multimedia tools.
  Interventions: Behavioral: Mental Health CPR
- Standard Community Health Education (Active Comparator): Participants in this arm receive standard community health education about mental health and wellness, without the structured Mental Health CPR behavioral components. This comparator arm allows for the evaluation of the added benefit of the Mental Health CPR intervention beyond general health education. Due to ethical considerations, the community-led intervention will be offered to the control arm after the community-intervention arm is completed. Participants in this arm will receive standard community health education materials about mental health and wellness, without the Mental Health CPR behavioral training components. This serves as the comparison group to evaluate the effectiveness of the intervention.
  Interventions: Behavioral: Standard Community Health Education

INTERVENTIONS:
Behavioral: Mental Health CPR — The Mental Health CPR is a culturally adapted behavioral intervention implemented by trained Community Mental Health Workers (CMHWs). It includes interactive sessions designed to improve emotional well-being, communication between cancer survivors and caregivers, and access to mental health services. The content integrates educational videos, group discussions, and digital resources from the Community Mental Health Toolbox. The intervention also reinforces sustainability by promoting local resource use and peer support networks. Additionally, the intervention will periodically conduct mental health and distress screenings, integrate mental health promotion educational activities and skill-building activities, case management component will integrate the cancer-mental health toolbox and linkage to Psycho-Oncology Mental Health Services (MHCS) component through the PAPSI psycho-oncology mental health service program at PHSU if needed.
  Arms: Mental Health CPR Intervention
Behavioral: Standard Community Health Education — The control group receives standard behavioral health education materials commonly distributed in community health settings. These materials include information on stress reduction, healthy lifestyle habits, and general mental health awareness but do not include interactive or CMHW-facilitated sessions.
  Arms: Standard Community Health Education

SUMMARY:
This is a parallel, two-arm interventional study comparing the Mental Health CPR behavioral intervention to standard community health education. The goal of this clinical trial is to learn if Mental Health CPR program, a culturally and linguistically adapted behavioral intervention, helps improve emotional well-being and access to mental health services among Hispanic/Latino cancer survivors in Puerto Rico.

The main questions it aims to answer are:

* Does Mental Health CPR help more people complete psychological distress screening?
* Does it help more participants connect with psycho-oncology services? Researchers will compare the Mental Health CPR program to standard community health education to determine whether it improves emotional well-being, enhances communication between patients and caregivers, reduces negative attitudes toward mental health care, and lowers emotional distress levels.

Participants will:

* Attend community sessions led by trained Community Mental Health Workers (CMHWs)
* Receive printed materials and educational resources
* Take part in brief follow-ups over about 36 weeks

DETAILED DESCRIPTION:
Mental Health CPR is a community-based behavioral intervention designed to improve access to psycho-oncology care and promote psychological well-being among Hispanic/Latino cancer survivors in Puerto Rico. The program was developed through a community-engaged process to ensure cultural and linguistic appropriateness and sustainability.

The study employs a cluster randomized parallel design in which community clusters are assigned to one of two conditions: the Mental Health CPR intervention or a standard community health education program. Trained Community Mental Health Workers (CMHWs) implement both arms concurrently over a 36-week period.

The Mental Health CPR intervention includes:

* Multimedia community sessions addressing emotional health and coping after cancer;
* Printed educational materials on distress screening and mental health resources; and
* Follow-up to reinforce key messages and promote connection to psycho-oncology services.

The comparison attention control group will be invited to attend general health fairs in which mental health printed educational materials will be available along with distress screening assessment.

Primary outcomes include completion of distress screening and uptake of psycho-oncology services. Secondary outcomes assess emotional distress, patient-caregiver communication, attitudes toward mental health care, quality of life, resilience, and selected salivary biomarkers related to stress and inflammation.

The study's findings will inform future strategies to enhance access to psycho-oncology services, strengthen the capacity of community-based health workers, and promote mental health care among cancer survivors living in under-supported communities.

ELIGIBILITY:
The study will include adults of all ages representing individuals across all the adulthood stage. The minimum age requirement is 21, which is the legal age of majority in Puerto Rico.

Inclusion Criteria:

* Eligibility Criteria for Sub-Aim 1a. The eligibility criteria for the qualitative interviews will be 1: Participants over 21 years old, 2: through their role or status, represent any of the following community sectors: cancer care community organization representatives, clinical care providers of cancer patients and survivors, and cancer health educators; 3: self-identified as a Latino/Hispanic; 4: be able to complete an interview.
* Eligibility Criteria for Aim 2. Community Forums stakeholders eligibility criteria. The community stakeholders inclusion criteria for the community forum are 1: Participants over 21 years old, 2: through their role or status, represent any of the following community sectors: cancer patients/survivors, cancer patients/survivors identified family caregiver, healthcare providers, cancer supportive care organizations, and advocacy groups, 3: self-identified as a Latino/Hispanic, 4: be able to attend the community forums.
* Community Leaders Eligibility Criteria for CMHW training. The inclusion criteria for the community leaders to be trained as CMHW are 1: Participants over 21 years of age, 2: living in a limited resource community in southern Puerto Rico, 3: self-identified as a Latino/Hispanic, and 4: be able to provide support to H-CAPS through their role as CMHW.
* Communities Eligibility Criteria. Community municipalities included from the southern health region of Puerto Rico are: Ponce, Arroyo, Coamo, Yauco, Salinas, Guanica, Guayanilla, Juana Diaz, Adjuntas, Guayama, Patillas, Santa Isabel, Penuelas and Villalba. These municipalities were chosen because they represent the catchment area of Ponce Health Sciences University.

Also, they are comprised of mostly rural areas (south-central region of Puerto Rico) and present a higher incidence of cancer (south region) and cancer mortality (south-central region) compared to other Puerto Rican Health regions.

* Intervention eligibility criteria. The eligibility criteria for the community intervention are 1: Participants over 21 years old, 2: living in any of the municipalities of the southern health region of Puerto Rico and within a limited resource community according to the CDC SVI, 3: self-identified as a Latino/Hispanic, and 4: have had a cancer diagnosis during their adulthood.

Exclusion Criteria:

* Participants residing outside the catchment area.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Development of the Community Toolbox for the Mental Health CPR Intervention | 18 months
  This outcome reflects the successful design, adaptation, and completion of the Community Toolbox - a culturally and linguistically tailored set of multimedia and printed resources developed to support the implementation of the Mental Health CPR intervention by Community Mental Health Workers (CMHWs). The Toolbox integrates educational modules, testimonial videos, infographics, and text message templates addressing distress screening, stigma reduction, communication enhancement, and linkage to psycho-oncology services. Completion is defined as finalization of all Toolbox modules validated through expert and community stakeholder review under Specific Aim 1.
Distress Thermometer (DT) | 9 months
  The Distress Thermometer (DT) is a validated single-item visual analog screening tool developed by the National Comprehensive Cancer Network (NCCN) to measure psychological distress in cancer patients. Participants rate their distress over the past week on a scale from 0 (no distress) to 10 (extreme distress). Higher scores indicate greater emotional distress. Mean DT score (0-10 scale)
Psych-oncology mental health service referral uptake | 9 months
  The percentage of participants who, after being screened for psychological distress, accept and complete at least one referral to psycho-oncology or behavioral health services. Uptake will be defined as documented attendance at one or more sessions with a licensed mental health or psycho-oncology provider. Data will be collected through Community Mental Health Worker (CMHW) tracking logs and verified by participant follow-up. Higher percentages indicate greater engagement in mental health services following the intervention.

SECONDARY OUTCOMES:
Communication and Caregiving Assessment Tool (Patient Form - CCAT-PF) | 9 months
  The Communication and Caregiving Assessment Tool - Patient Form (CCAT-PF) is a validated self-report scale that assesses the quality and effectiveness of communication between patients and their primary caregivers. The scale includes items rated on a Likert-type format to evaluate understanding, emotional support, and problem-solving aspects of the patient-caregiver relationship. Higher scores indicate better communication quality. Mean score on the CCAT-PF (range 1-5)
Communication and Caregiving Assessment Tool (Caregiver Form - CCAT-CF) | 9months
  The Communication and Caregiving Assessment Tool - Patient Form (CCAT-PF) is a validated self-report instrument that measures the patient's perception of communication quality with their primary caregiver. Items are rated on a Likert-type scale assessing emotional support, understanding, and collaborative problem solving. Higher scores indicate better communication quality. Mean CCAT-PF total score (range 1-5)
Self-Stigma of Mental Illness Scale (SSMIS) | 9 months
  The Self-Stigma of Mental Illness Scale (SSMIS), developed by Corrigan et al. (2006), is a validated 40-item self-report instrument that measures internalized stigma toward mental illness and help-seeking. The SSMIS assesses four sequential components of self-stigma: awareness of stereotypes, agreement with stereotypes, application of stereotypes to oneself, and harm to self-esteem. Items are rated on a 9-point Likert scale (1 = strongly disagree to 9 = strongly agree). Higher scores indicate greater self-stigma. Mean SSMIS total score (range 1-9)
Psychological distress, assessed with the Hospital Anxiety and Depression Scale (HADS) | 9 months
  The Hospital Anxiety and Depression Scale (HADS), is a validated 14-item self-report questionnaire designed to assess symptoms of anxiety and depression in medical and community populations. It consists of two subscales-HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D)-each containing 7 items scored from 0 to 3. Subscale scores range from 0 to 21, with higher scores indicating greater anxiety or depression symptom severity. Mean HADS-A and HADS-D subscale scores (range 0-21)
Health-Related Quality of Life assessed with the Functional Assessment of Cancer Therapy - General (FACT-G, Version 4) | 9 months
  The Functional Assessment of Cancer Therapy - General (FACT-G, Version 4) is a validated 27-item questionnaire developed by Cella et al. (1993) that measures health-related quality of life in cancer patients across four domains: Physical, Social/Family, Emotional, and Functional Well-Being. Each item is rated on a 5-point Likert-type scale (0-4). Higher scores indicate better quality of life.
  Population: Adult cancer survivors enrolled in the Mental Health CPR study. Unit of Measure: Mean FACT-G total score (range 0-108)
Perceived Social Support, asses with Multidimensional Scale of Perceived Social Support (MSPSS) | 9 months
  The Multidimensional Scale of Perceived Social Support (MSPSS), developed by Zimet et al. (1988), is a validated 12-item self-report questionnaire that measures perceived social support from three sources: family, friends, and significant others. Each item is rated on a 7-point Likert scale (1 = very strongly disagree to 7 = very strongly agree). Higher total scores indicate greater perceived social support. Mean MSPSS total score (range 1-7)
Brief Resilience Scale (BRS) | 9 months
  The Brief Resilience Scale (BRS), developed by Smith et al. (2008), is a 6-item self-report questionnaire designed to assess the ability to recover from stress. Items are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Higher scores reflect greater resilience. Mean BRS total score (range 1-5)
Salivary Stress Hormone Levels (Cortisol and Alpha-Amylase) | 9 months
  Salivary cortisol and alpha-amylase levels will be measured as biomarkers of physiological stress response. Saliva samples will be collected from participants at baseline and post-intervention following standardized collection procedures (e.g., morning fasting samples). Samples will be stored and analyzed in a blinded laboratory setting using enzyme-linked immunosorbent assay (ELISA) and kinetic enzyme assays. Higher cortisol and alpha-amylase concentrations indicate higher physiological stress activation. Laboratory personnel conducting assays are blinded to participants' group assignments. Mean salivary cortisol (µg/dL); mean salivary alpha-amylase (U/mL)
Salivary Cytokine and Chemokine Concentrations | 9 months
  Salivary cytokine and chemokine concentrations will be analyzed as biomarkers of inflammation and immune activation associated with stress response. Samples will be collected using standardized saliva collection procedures and stored at -80°C until analysis. Laboratory assays will be performed using multiplex immunoassay or enzyme-linked immunosorbent assay (ELISA) methods to quantify cytokines (e.g., IL-6, IL-10, TNF-α) and chemokines (e.g., MCP-1, IL-8). All laboratory personnel conducting the analyses are blinded to participants' group assignments to ensure unbiased outcome assessment. Higher concentrations reflect greater inflammatory response. Mean concentration (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Eida M Castro-Figuera, PsyD, MSc, Principal Investigator — Ponce Medical School Foundation, Inc.
Locations (1):
- Ponce Medical School Foundation, Inc., Ponce, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data, data dictionary, and supporting documentation will be deposited in a Trans-NIH BMIC-approved generalist repository following publication of the primary results. Data will be curated under FAIR principles and protected under a Certificate of Confidentiality.
Time Frame: All data gathered by this research will be publicly available no later than publication acceptance of the main findings